CLINICAL TRIAL: NCT06982638
Title: Accelerated TMS for Freezing of Gait in Parkinson's Disease
Acronym: TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Gonzalo Revuelta, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00138900
Record Dates: First submitted 2025-04-23; First posted 2025-05-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD)
Keywords: TMS; Parkinson's Disease (PD); Gait training; Freezing of gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TMS+Gait training (Experimental): Participants in this single-arm study will receive a personalized, accelerated course of continuous theta burst stimulation (cTBS) over a functionally defined subregion of the supplementary motor area (SMA), which is individually targeted using resting-state functional MRI. The stimulation will be delivered using a MagPro Cool-B65 A/P figure-of-eight coil at 110% of resting motor threshold.
  Each participant will undergo 6 treatment visits over 2 weeks , receiving 8 rTMS sessions per day (600 pulses/session), totaling 28,800 pulses across the study. TMS sessions will be interleaved with dual-task gait training involving cognitive walking exercises. Gait training will be conducted for 30 minutes per visit, immediately following stimulation blocks. Safety, tolerability, adherence, gait performance, and neuroplasticity will be evaluated pre- and post-intervention using clinical scales, motor evoked potentials (MEPs), and functional MRI.
  Interventions: Device: TMS+ Gait training

INTERVENTIONS:
Device: TMS+ Gait training — Participants in this single-arm study will receive a personalized, accelerated course of continuous theta burst stimulation (cTBS) over a functionally defined subregion of the supplementary motor area (SMA), which is individually targeted using resting-state functional MRI. The stimulation will be delivered using a MagPro Cool-B65 A/P figure-of-eight coil at 110% of resting motor threshold.
  Each participant will undergo 6 treatment visits over 2 weeks , receiving 8 rTMS sessions per day (600 pulses/session), totaling 28,800 pulses across the study. TMS sessions will be interleaved with dual-task gait training involving cognitive walking exercises. Gait training will be conducted for 30 minutes per visit, immediately following stimulation blocks. Safety, tolerability, adherence, gait performance, and neuroplasticity will be evaluated pre- and post-intervention using clinical scales, motor evoked potentials (MEPs), and functional MRI.

SUMMARY:
The goal of this clinical trial is to learn whether a personalized brain stimulation method called repetitive transcranial magnetic stimulation (rTMS), combined with walking exercises, is a practical and tolerable approach to help people with Parkinson's disease who experience freezing of gait (FOG). FOG is a disabling symptom where people temporarily feel stuck and unable to start walking, even though they want to move.

The main questions this study aims to answer are:

Can people with Parkinson's disease and FOG tolerate this combined rTMS and walking training procedure?

Can researchers successfully enroll and retain participants for this multi-visit intervention?

Does the combination of rTMS and gait training show early signs of improving gait and reducing freezing episodes?

This study does not include a comparison or placebo group. All participants will receive the same intervention.

Participants will:

Attend up to 15 study visits over about 16 weeks, with the option to combine visits to reduce burden.

Complete brain imaging (MRI) before and after the intervention to guide and evaluate treatment.

Receive a form of brain stimulation (rTMS) using a safe, non-invasive coil placed over a specific part of the brain called the supplementary motor area (SMA). The target is personalized using each person's MRI data.

Participate in walking exercises that include cognitive tasks (dual-task gait training) after each set of brain stimulation sessions.

Undergo assessments of walking ability, Parkinson's disease symptoms, and brain response to stimulation.

Be videotaped during walking tasks to assess gait changes, while wearing small motion sensors on the body.

Complete questionnaires about symptoms, safety, and tolerability.

This study is being conducted at the Medical University of South Carolina (MUSC) and includes up to 15 adults between the ages of 50 and 80 who have been diagnosed with Parkinson's disease and experience FOG.

Although rTMS is already FDA-cleared for depression and other conditions, it has not been approved for freezing of gait, and its use in this study is considered investigational. The stimulation device used has been determined to be non-significant risk (NSR) by the FDA.

The study does not offer direct medical benefit to participants, but results from this trial may help researchers develop future treatments and better understand how brain stimulation affects walking difficulties in Parkinson's disease.

Participation is voluntary, and individuals can withdraw from the study at any time without affecting their medical care

ELIGIBILITY:
Inclusion Criteria:

1. 50-80 years of age
2. diagnosis of PD based on UK Brain Bank diagnostic criteria 55
3. presence of FOG defined as a score of 1 on part 1 of the nFOGQ in which a video showing different types of freezing is played for the patient, a score of 1 represents a positive response of having experienced such an episode over the last month
4. no dopaminergic medication changes in the month prior
5. observed FOG rated as >1 in item 3.11 of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

Exclusion Criteria:

1. a history of other significant gait impairment unrelated to PD (e.g. orthopedic deformities)
2. inability to complete gait assessments (timed up and go task) without assistance or assist devices
3. barriers to making contact between the TMS coil and the skin (e.g. braids that cannot be removed)
4. failing to meet all criteria on a standardized MRI/TMS safety screening: This includes, but is not limited to, the presence of claustrophobia, implanted electronic devices (e.g., pacemakers), metallic objects or fragments (e.g., bullets), and non-removable hair clips or piercings.
5. individuals with a diagnosis of psychosis or any other cognitive impairments that would make them unable to understand and follow study instructions or to consent for themselves.
6. pregnancy
7. individuals with a history of seizure

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerability of the Intervention | Immediately after each TMS session during the 6 treatment days
  Participant-reported discomfort after each TMS session using a modified version of the Non-Invasive Brain Stimulation (NIBS) Tolerability Questionnaire, which rates six side effects (headache, pain, scalp irritation, facial twitching, fatigue, fear/anxiety) from 1 (Mild) to 10 (Severe).
Adherence to Study Visits | Across the total study duration, up to 16 weeks
  The proportion of scheduled study visits completed by each participant, calculated as the number of attended sessions divided by the number of planned sessions.

SECONDARY OUTCOMES:
Change in Freezing of Gait Questionnaire Scores (nFOG-Q) | nFOG-Q will be assessed at 5 time points: 1)Baseline 2) immediately after completion of intervention 3) one month after completion of intervention, 4)two months after completion of intervention 5) three months after completion of intervention
  Difference in participant-reported FOG severity using the New Freezing of Gait Questionnaire (nFOG-Q) from baseline to post-intervention.
Change in MDS-UPDRS Gait Item Scores | Baseline and after completion of intervention, up to 16 weeks
  Changes in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) gait-related items, especially item 3.11 (FOG), assessed before and after the intervention.
Change in SMA Functional Connectivity | Baseline and after completion of intervention, up to 16 weeks
  Pre-to-post change in resting-state fMRI connectivity between the supplementary motor area (SMA) and other brain regions, particularly the cerebellar locomotor region (CLR).

OTHER OUTCOMES:
Cortical Plasticity via MEP Amplitude Changes | Baseline
  Change in motor evoked potential (MEP) amplitude following administration of continuous and intermittent theta burst stimulation (cTBS and iTBS) over the motor cortex, measured at 0, 5, 10, 15, 20, and 30 minutes post-stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carlina, Charleston, South Carolina, United States